CLINICAL TRIAL: NCT05511025
Title: A Phase I Randomized Single-blind Placebo-controlled Study to Assess the Safety, Tolerability, and Pharmacokinetics of AZD6234 Following Single Ascending Dose Administration to Healthy Subjects Who Are Overweight or Obese
Brief Title: Assess the Safety, Tolerability, and Pharmacokinetics of AZD6234 Following Single Ascending Dose Administration to Healthy Subjects Who Are Overweight or Obese
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: D8750C00001
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Healthy Participants
Keywords: Overweight; Obese; Non-childbearing
MeSH Terms: conditions — Overweight; Obesity | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1 (Experimental): Participants will receive single ascending doses of AZD6234 via SC injection and matching volumes of the placebo as a solution via SC
  Interventions: Drug: AZD6234; Drug: Placebo; Combination Product: Acetaminophen
- Cohort 2 (Experimental): Participants will receive a single dose of AZD6234 via an SC injection and matching volume of the placebo as a solution via SC injection
  Interventions: Drug: AZD6234; Drug: Placebo; Combination Product: Acetaminophen
- Cohort 3 (Experimental): Participants will receive single ascending doses of AZD6234 via SC injection and matching volumes of the placebo as a solution via SC injection
  Interventions: Drug: AZD6234; Drug: Placebo; Combination Product: Acetaminophen
- Cohort 4 (Experimental): Participants will receive single ascending doses of AZD6234 via IV injection and matching volumes of the placebo as a solution via IV injection
  Interventions: Drug: AZD6234; Drug: Placebo; Combination Product: Acetaminophen
- Cohort 5 (Experimental): One dose level for SC administration is planned to be investigated for Japanese participants only
  Interventions: Drug: AZD6234; Drug: Placebo; Combination Product: Acetaminophen
- Cohort 6 (Experimental): Participants will receive single ascending doses of AZD6234 via SC injection and matching volumes of the placebo as a solution via SC injection
  Interventions: Drug: AZD6234; Drug: Placebo; Combination Product: Acetaminophen
- Cohort 7 (Experimental): Participants will receive single ascending doses of AZD6234 via SC injection and matching volumes of the placebo as a solution via SC injection
  Interventions: Drug: AZD6234; Drug: Placebo; Combination Product: Acetaminophen
- Cohort 8 (Experimental): Participants will receive AZD6234 via SC injection and matching volumes of placebo as a solution via SC injection
  Interventions: Drug: AZD6234; Drug: Placebo; Combination Product: Acetaminophen

INTERVENTIONS:
Drug: AZD6234 — Participants will receive a single dose of AZD6234 as a solution via SC or IV injection
Drug: Placebo — Participants will receive matching volumes of the placebo as a solution via SC or IV injection
Combination Product: Acetaminophen — Participants will receive a single dose of acetaminophen as part of a meal

SUMMARY:
A study in healthy male and female participants of non-childbearing potential who are overweight or obese.

DETAILED DESCRIPTION:
The study will comprise of:

* A Screening Period of maximum 28 days.
* A Treatment Period during which participants will be resident at the Clinical Unit from three days before (Day -3 ) Investigational Medicinal Product (IMP) administration (Day 1) until at least 4 days (96 hours) after IMP administration, participants will then be discharged on the morning of Day 5.
* Weekly outpatient visits on Days 8, 15, 22, 29, and 36 for blood sample collection, Electrocardiogram (ECGs), and adverse events (AE) recording.
* A Follow-up Visit 6 weeks (Day 43) after the last IMP dose.

Furthermore, 3 dose levels of AZD6234 for Subcutaneous (SC) administration (Cohorts 1 to 3) and one dose level for Intravenous (IV) administration (Cohort 4) are planned to be investigated in healthy participants who are overweight or obese. The IV cohort (Cohort 4) can begin in parallel or after Cohort 3. One dose level for SC administration is planned to be investigated in Japanese participants only (Cohort 5), and up to 3 additional dose levels for SC administration are planned to be investigated in healthy participants (Cohort 6 to 8). Depending on the findings, additional (optional) dose level cohorts may be added at the discretion of the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Healthy male and female participants aged 18 to 55 years with suitable veins for cannulation or repeated venipuncture.
* Females must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit, must not be lactating and must be of non childbearing potential, confirmed at the Screening Visit by fulfilling one of the following criteria:

  (i) Post menopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and Follicle stimulating hormone (FSH) levels in the post menopausal range.

(ii) Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.

* Have a body mass index (BMI) of 25 to 35 kg/m2 inclusive (at the time of screening) and weigh at least 50 kg.

For the Japanese cohort(s):

* Participant is a native of Japan; defined as having both parents and four grandparents who are Japanese. This includes second and third generation subjects of Japanese descent whose parents or grandparents are living in a country other than Japan.
* Have a BMI of 23 to 35 kg/m2 inclusive (at the time of screening) and weigh at least 50 kg.

Exclusion Criteria:

* History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study, including:

  (i) Gastroparesis (or similar) requiring treatment, or (ii) Previous surgery of the upper gastrointestinal tract, or (iii) Cardiovascular disease, including but not limited to sick sinus syndrome, valvular disease, and cardiomyopathy, or (iv) Neuromuscular or neurogenic disease, or (v) Severe vitamin D deficiency < 12 ng/dL (as assessed by screening laboratory results or history), or (vi) Type 1 or type 2 diabetes mellitus.
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
* Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IMP.
* Any laboratory values with the following deviations:

  (i) Alanine aminotransferase > Upper limit of normal (ULN) (ii) Aspartate aminotransferase > ULN (iii) eGFR < 60 ml/min/1.73 m2 (calculated using the CKD EPI formula) (iv) White blood cell count < LLN (v) Hemoglobin < LLN (vi) Total calcium or corrected calcium/ionized calcium < LLN or > ULN
* Abnormal vital signs, after 10 minutes supine rest, defined as any of the following:

  (i) Systolic Blood pressure (BP) < 90 mmHg or > 140 mmHg. (ii) Diastolic BP < 50 mmHg or > 90 mmHg. (iii) Heart rate < 55 or > 85 beats per minute (bpm)
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD6234.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within at least 30 days or 5 half-lives (whichever is longer) of the first administration of IMP in this study. The period of exclusion begins 30 days or 5 half-lives after the last visit in the previous study, whichever is the longest.
* Participants who are vegans or have medical dietary restrictions.
* Vulnerable participants, eg, kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with AEs and Serious Adverse Events(SAE) | From Screening until Follow up (Day 43)
  The safety and tolerability of AZD6234 following subcutaneous and/or intravenous administration of single ascending doses in healthy participants, including Japanese participants, who are overweight or obese will be assessed.

SECONDARY OUTCOMES:
Maximum observed plasma drug concentration (Cmax) | From Day 1 until Follow up (Day 43)
  The pharmacokinetics of AZD6234 in plasma following subcutaneous and/or intravenous administration of single ascending doses of AZD6234 in healthy participants, including Japanese participants, who are overweight or obese will be assessed.
Area under the plasma concentration-time (AUClast) | From Day 1 until Follow up (Day 43)
  The pharmacokinetics of AZD6234 in plasma following subcutaneous and/or intravenous administration of single ascending doses of AZD6234 in healthy participants, including Japanese participants, who are overweight or obese will be assessed.
Area under plasma concentration-time curve from zero to infinity (AUCinf) | From Day 1 until Follow up (Day 43)
  The pharmacokinetics of AZD6234 in plasma following subcutaneous and/or intravenous administration of single ascending doses of AZD6234 in healthy participants, including Japanese participants, who are overweight or obese will be assessed.
Time to reach maximum observed concentration (tmax) | From Day 1 until Follow up (Day 43)
  The pharmacokinetics of AZD6234 in plasma following subcutaneous and/or intravenous administration of single ascending doses of AZD6234 in healthy participants, including Japanese participants, who are overweight or obese will be assessed.
Terminal rate constant (λz) | From Day 1 until Follow up (Day 43)
  The pharmacokinetics of AZD6234 in plasma following subcutaneous and/or intravenous administration of single ascending doses of AZD6234 in healthy participants, including Japanese participants, who are overweight or obese will be assessed.
Terminal elimination half-life (t½λz) | From Day 1 until Follow up (Day 43)
  The pharmacokinetics of AZD6234 in plasma following subcutaneous and/or intravenous administration of single ascending doses of AZD6234 in healthy participants, including Japanese participants, who are overweight or obese will be assessed.
Total body clearance of drug from plasma (IV dosing only) (CL) | From Day 1 until Follow up (Day 43)
  The pharmacokinetics of AZD6234 in plasma following subcutaneous and/or intravenous administration of single ascending doses of AZD6234 in healthy participants, including Japanese participants, who are overweight or obese will be assessed.
Apparent total body clearance of drug from plasma (SC dosing only) (CL/F) | From Day 1 until Follow up (Day 43)
  The pharmacokinetics of AZD6234 in plasma following subcutaneous and/or intravenous administration of single ascending doses of AZD6234 in healthy participants, including Japanese participants, who are overweight or obese will be assessed.
Volume of distribution based on the terminal phase (IV dosing only) (Vz) | From Day 1 until Follow up (Day 43)
  The pharmacokinetics of AZD6234 in plasma following subcutaneous and/or intravenous administration of single ascending doses of AZD6234 in healthy participants, including Japanese participants, who are overweight or obese will be assessed.
Apparent volume of distribution based on the terminal phase (SC dosing only) (Vz/F) | From Day 1 until Follow up (Day 43)
  The pharmacokinetics of AZD6234 in plasma following subcutaneous and/or intravenous administration of single ascending doses of AZD6234 in healthy participants, including Japanese participants, who are overweight or obese will be assessed.
Dose-normalized AUClast (AUClast/D) | From Day 1 until Follow up (Day 43)
  The pharmacokinetics of AZD6234 in plasma following subcutaneous and/or intravenous administration of single ascending doses of AZD6234 in healthy participants, including Japanese participants, who are overweight or obese will be assessed.
Dose-normalized AUCinf (AUCinf/D) | From Day 1 until Follow up (Day 43)
  The pharmacokinetics of AZD6234 in plasma following subcutaneous and/or intravenous administration of single ascending doses of AZD6234 in healthy participants, including Japanese participants, who are overweight or obese will be assessed.
Dose-normalized Cmax (Cmax/D) | From Day 1 until Follow up (Day 43)
  The pharmacokinetics of AZD6234 in plasma following subcutaneous and/or intravenous administration of single ascending doses of AZD6234 in healthy participants, including Japanese participants, who are overweight or obese will be assessed.
Time of last observed (quantifiable) concentration (tlast) | From Day 1 until Follow up (Day 43)
  The pharmacokinetics of AZD6234 in plasma following subcutaneous and/or intravenous administration of single ascending doses of AZD6234 in healthy participants, including Japanese participants, who are overweight or obese will be assessed.
Prevalence and incidence of anti-drug antibodies (ADAs) to AZD6234 | Day 1, Day 15, Day 29 and at Follow up (Day 43)
  The immunogenicity following subcutaneous and/or intravenous administration of single ascending doses of AZD6234 in healthy participants, including Japanese participants, who are overweight or obese will be assessed.
ADA titer | Day 1, Day 15, Day 29 and at Follow up (Day 43)
  The immunogenicity following subcutaneous and/or intravenous administration of single ascending doses of AZD6234 in healthy subjects, including Japanese subjects, who are overweight or obese will be assessed

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Research Site, Glendale, California
  - Research Site, Brooklyn, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home